# Characteristics of Balance Control to Unexpected Loss of Balance During Standing and Walking in Post-stroke Individuals

#NCT02619175

Date: 09.02.2019

# **Protocol**

# **Participants**

PwS were recruited during their hospitalization at the Loewenstein Rehabilitation Hospital (LRH), Ra'anana, Israel between November 2016 to February 2018. Inclusion criteria included first unilateral stroke, being able to walk with or without a walking aid independently or under supervision. Exclusion criteria included body weight greater than 135 kg, other neurological disorders, severe arthritis, joint replacement surgery and blindness, confirmed by the individuals' physician and medical record at the time of enrollment. The study was approved by the Institutional Review Board at the Loewenstein Hospital (approval number LOE-14-0021). Participants signed a written informed consent according to the declaration of Helsinki.

# Study design

Subacute PwS were randomized to perturbation-based balance training (PBBT) or weight shifting and gait training (WS&GT). Allocation was made by an investigator not involved in the assessments using computer random allocation software (Random Allocation Software Version 1.1, Isfahan Iran). Participants were tested before and after the training period by a blinded investigator. PwS in the PBBT and WS&GT groups received 12 training sessions, each session lasted 30 minutes, 1 training session per day over a period of 2.5 weeks. Pretraining (T1) and post training (T2) assessments included laboratory reactive balance capacity functions and clinical measures of balance, gait, motor impairments, and balance confidence. Follow-up assessment (T3) conducted 5 weeks after intervention completion and included only assessment of reactive balance capacity. All assessment sessions were performed at the same time of day and in the same order.

# <u>Assessment Protocol</u>

Participants stood on a computerized mechatronic treadmill system that provides unannounced perturbations by a horizontal movable platform (Balance Tutor, MediTouch Ltd, Israel), wearing a safety harness that prevented falls but did not

restrict their movements. Surface translations were increased systematically in 6 intensities from low (intensity 1) to high (intensity 6) for a total of 24 perturbation trials (characteristics of perturbation intensities are described in Table 1).. Participants were instructed to stand with feet placed together and to react naturally to prevent themselves from falling. A safety harness system was attached to an overhead track via rope. Rope length was adjusted individually so it would prevent participants' knees from touching the treadmill belt in case of fall. In case of a fall into harness, the participant did not continue to higher intensity. Participants performed all trials wearing their own sport shoes and foot orthosis in case they needed ankle support.

### **Outcome measures**

Reactive balance capacity was assessed by multiple-step threshold and fall threshold. Multiple-step threshold was defined as the minimum perturbation intensity that consistently elicits 2 or more compensatory steps that extended the base of support in at least 2 consecutive perturbation intensities. Fall threshold was defined as the perturbation intensity that results in unsuccessful balance recovery, that is, when a subject was unambiguously supported by the harness system. Multiple-step threshold and fall threshold have been found to demonstrate high interrater and test retest reliability in healthy adults. In case a participant did not fall at the highest perturbation intensity (intensity 6), his or her fall threshold was calculated as intensity 7. Reactive step initiation time, step length and step velocity were measured using a three-dimensional motion analysis system (APAS inc).

A day prior to the reactive balance assessment, PwS underwent a clinical assessment that included the lower extremity Fugl-Meyer (LEFM) assessment, Berg Balance Scale (BBS), 10-meter walk test (10MWT), 6-minute walk test (6MWT), and Activity-specific Balance Confidence (ABC) scale. These measures have been found to demonstrate strong interrater and test-retest reliability in PwS.

### **Intervention Programs**

### Group 1 - Perturbations based balance training

In the PBBT group, each training session consisted of 36 random right/left/forward/backward unannounced platform translations while standing (i.e. 3 blocks of 12 perturbations) and 30 random right/left perturbations during a 10- to 12-minute treadmill walk (Balance Tutor, MediTouch Ltd, Israel). Perturbations were synchronized to the single support phase of gait cycle using the Balance Tutors' inertial sensors. Perturbations were unpredicted in terms of time and direction. The instruction was "try to prevent yourself from falling." In the first training session, the initial perturbation intensity was individually adjusted according to participant's maximal ability, that is, the maximal perturbation intensity that could be recovered without falling into harness system during the baseline assessment. Progression to higher intensity occurred if the participant was able to recover from 24 consecutive perturbations (2 blocks of 12 perturbations) without a fall and felt that he or she could be further challenged. The increase in intensity during training was constant and a function of the following perturbation parameters: in forward and backward perturbations: distance = 1.86 cm, velocity = 3.65 cm/s, and acceleration = 11.72 cm/s2 and in response to lateral perturbations: distance = 1.17 cm, velocity = 3.79 cm/s, and acceleration = 12.07 cm/s2.

## Group 2 – Weight shifting and gait training (control)

In the WS&GT group, each session consisted of 36 voluntary weight shifting exercises (3 blocks of 12 targets) delivered in a random order while standing on a computerized force platform (Balance Master, NeuroCom International Inc) and a 10- to 12-minute treadmill walk without perturbations. For weight shifting, participants stood on a force platform while viewing a display of their center of pressure position relative to a target on a screen. They were instructed to shift weight in order to reach the target without changing their feet position or falling. In the first session, the initial distance for weight shifting was individually adjusted for each participant as the maximal distance he or she could shift weight without falling into harness or changing their feet position. The distance to target was increased by 5% if the participant was able to complete a set of 24 consecutive

weight siftings without falling or changing their feet position and felt that he or she could be further challenged (Figure 2). Participants in both groups walked at their preferred treadmill walking speed that was adjusted during sessions according to their abilities. In case the participants needed, support was given by the therapist's hand. To increase task difficulty in both groups a concurrent cognitive task was added (backward counting by 3 or 7) in training sessions 9 to 12. Participants were provided information regarding knowledge of the results of the balance reaction, that is, the occurrence of a fall into harness, through information inherent in the task (the pull of the harness) and verbal feedback regarding perturbation intensity/weight shifting distance and walking speed. At the end of each session participants were asked to rate their perceived level of challenge on a 0-to-10 scale where 0 represents no challenge and 10 represents very high challenge. During the study period, PwS continued with their regular rehabilitation therapies that included daily physical therapy and occupational therapy treatments and if needed, speech therapy treatment. All measurement and training sessions were conducted by physical therapists working in neurological rehabilitation.

### Statistical analyses

Baseline characteristics will be compared using independent-samples t test for continuous variables, Mann-Whitney U test for ordinal variables or variables with non-normal distributions, and chi-square test for categorical data. A mixed factorial analysis of variance for normally distributed dependent variables will be conducted. The independent variables are group (PBBT, WS&GT) and time (baselineT1, postintervention-T2, follow-up-T3). In case of non-normal distributions or ordinal variables the Mann-Whitney U test will be used to compare group-by-time interactions by computing the differences between post intervention and baseline performances (T2-T1) and between follow-up and baseline performances (T3-T1).

Table 1. Perturbation parameters by perturbation intensity and direction.

| Perturbation | Forwa | rd/Backwa | rd surface | Rightward/Leftward surface translation | | |
|---|---|---|---|---|---|---|
| Intensity | | translatio | on | | | |
| | Distance | Velocity | Acceleration | Distance | Velocity | Acceleration |
| | (cm) | (cm/sec) | (cm/sec <sup>2</sup> ) | (cm) | (cm/sec) | (cm/sec <sup>2</sup> ) |
| 1 | 10.44 | 17.62 | 126.89 | 5.68 | 20.17 | 73.27 |
| 2 | 14.17 | 24.93 | 150.34 | 8.03 | 27.75 | 97.41 |
| 3 | 17.89 | 32.24 | 173.79 | 10.37 | 35.34 | 121.55 |
| 4 | 21.62 | 39.55 | 197.24 | 12.72 | 42.93 | 145.68 |
| 5 | 25.34 | 46.86 | 220.69 | 15.06 | 50.51 | 169.82 |
| 6 | 29.06 | 54.17 | 244.13 | 17.41 | 58.10 | 193.96 |

Abbreviation: cm, centimetre; cm/sec, centimetre per second; cm/sec<sup>2</sup>, centimetre per second square.





# Berg Balance Scale (B.B.S.)

### <u>הנחיות:</u>

- המבחן כולל 14 משימות סטטיות ודינאמיות לשמירת שיווי משקל.
- כל משימה מקבלת ציון של 0 עד 4 נקודות- בהתאם לאיכות המשימה וזמן הביצוע.
  - ציון מירבי 56 נקודות.
  - בטופס המבחן קיימות הוראות לבצוע כל משימה בנפרד והציון לכל משימה.
    - בציון , נלקח בחשבון הביצוע הנמוד לכל משימה.
- ברוב המשימות הנבדק מתבקש לשמור על תנוחה מסויימת לאורך זמן. יש להוריד בציון אם הנבדק לא עומד בדרישת הזמן או המרחק המתבקש, או אם הנבדק נוגע בתמיכה חיצונית או נעזר בבודק.
- במשימות 8. (הושטת יד), 9. (הרמת חפץ מהקרקע) 13. (טנדם) ו-14. (עמידה על רגל אחת) הנבדק מחליט על רגל/יד.
- ציוד: סרגל עם סימון של 5,12,25 ס״מ, כסא סטנדרטי, בגובה סביר, מדרגה או שרפרף בגובה של מדרגה ממוצעת.



### References:

- 1) Berg et al, 1989
- 2) Berg et al, 1995
- 3) Walker et al, 2000
- 4) Steffen et al, 2002
- 5) Hatch et el, 2003
- 6) Salter et al, 2005
- 7) Australian Physiotherapy Association National Neurology Group, 2005





# Berg Balance Scale - מבחן שיווי משקל

| ם הנבדק: אבחנה | שכ |
|----------------|----|
|----------------|----|

| שיצה לעמידה: בבקשה קום לעמודה. נסה לא להשתמש ביחים לתמוכה מסוגול לעמוד ללא עורת ידיים ולהתייצב עצמאית מסוגול לעמוד לא עורת ידיים ולהתייצב עצמאית מסוגול לעמוד בעורת ידיים לאחר מסבר ניסיונות מסוגול לעמוד בעורת ידיים לאחר מסבר ניסיונות זיקול לעורה קבלית או מבדית לעמוד עמידה ללא תמיכה: עמוד במשך 2 דקות לא תמוכה מסוגול לעמוד בבטיחות 2 דקות מסוגול לעמוד בבטיחות 2 דקות מסוגול לעמוד במורת לעמוד 3 שניות ללא תמיכה מסוגול לעמוד מנות לעמוד 3 שניות ללא תמיכה מסוגול לעמוד מנות לא תמיכה משבת 2 בשילוב ידיים למשך 2 דקות אוני מוד לא תמיכה, רגליים על הרצמה: שב בשילוב ידיים למשך 2 דקות מסוגול לשבת במיחות למשך 3 דקות מסוגול לשבת במיחות למשך 3 דקות מסוגול לשבת במיחות למשך 3 דקות מסוגול לשבת במיחות למשך 3 דקות מסוגול לשבת מוד | תאריך<br>(3) | תאריך<br>(2) | תאריך<br>(1) | | |
|---|---|---|---|---|---|
| מסוגל לעמוד עצמאות בעורת ידיים לאחר מוסר ניסיונות מוסג לעמוד בעורת ידיים לאחר מוסר ניסיונות ודיים לאחר מוסר ניסיונות סומגל לעמוד בעורת ידיים לאחר מוסר ניסיונות עמידה ללא תמיכה: עמוד במשך 2 דקות ללא תמיכה מסוגל לעמוד בסיחות 2 דקות מסוגל לעמוד 2 דקות במשרחה מסוגל לעמוד 3 דקות במשרחה מסוגל לעמוד 3 דקות במשרחה מסוגל לעמוד 3 נשניות ללא תמיכה מסוגל לעמוד 3 נשניות ללא תמיכה ודיים ליסיונות לעמוד 3 נשניות ללא תמיכה מסוגל לעמוד 3 נשניות ללא תמיכה מסוגל לעמוד 3 נשניות ללא תמיכה מסוגל לעמוד 3 נשניות ללא מריכה מסוגל לעמוד 3 נשניות ללא מריכה מסוגל לשבת בבטיחות למשך 2 דקות מסוגל לשבת במיחות למשך 2 דקות מסוגל לשבת במיחות למשך 3 דקות מסוגל לשבת במיחות למשך 3 דקות מסוגל לשבת במיחות למשך 3 דקות מסוגל לשבת במיחות למשר מדיים מסוגל לשבת במיחות למשר מדיים מסוגל לשבת במיחות עם עזרה מינימלית של ידיים עולט בישיבה ע"י שימוש בידיים משתמש בנב הרגלים כנגד הכיסא לשליטה בישיבה משתמש בנב ברגלים כנגד הכיסא לשליטה בישיבה משתמש בנב ברגלים כנגד הכיסא למיטה ובחזרה. לכיוון כיסא עם משעות, ולכיוון כיסא ללא משעות משעמש בנב ביטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בטיחות עם עזרה מושית של ידיים מסוגל לעבור מידים עם עינים צומות יופנים את עיניך ועמוד ישר במשך 10 שניות עם הוא מושים מסוגל לעמוד 10 שניות במילה מסוגל לעמוד 10 שניות בסילה מסוגל לעמוד 10 שניות בסילה באום עצמאי לעמוד 1 דקה בבטיחות מסוגל לעמיד 10 שנית בלים באום עצמאי לעמוד 1 דקה בבטיחות מסוגל לעמיד רגליים באום עצמאי לעמוד 1 דקה בבטיחות מסוגל לעמיד רגליים באום עצמאי לעמוד 1 דקה בבטיחות מסוגל לעמיד רגליים באום ענמאי אך אינו מוסוגל לעמיד באום במיותות | | | | ישיבה לעמידה: בבקשה קום לעמידה. נסה לא להשתמש בידיים לתמיכה | 1 |
| מסוגל לעמוד בעורת ידיים לאחר מוסבר ניסיונות מוסבר לידים לאחר מוסבר ניסיונות מוסבר לידים לאור מיסבר מעמדה ללא תמיכה ועמוד בשור | | | | מסוגל לעמוד ללא עזרת ידיים ולהתייצב עצמאית | 4 |
| 1 זקוק לעזרה קלה לעמוד או להתייצב 2 עמידה ללא תמיכה: עמוד במשך 2 דקות ללא תמיכה 3 נסוגל לעמוד 2 דקות במשרח 2 דקות ללא תמיכה 3 מוטגל לעמוד 2 דקות במשרח 3 דקות למוטגל לעמוד 2 דקות במשרח 5 נסוגל לעמוד 2 דקות במשרח 6 מיסוגל לעמוד 3 דקות במשרח 6 מיסוגל לעמוד 3 דקות במשרח 6 מיסוגל לעמוד 3 דקות במשרח 5 מיסוגל לעמוד 3 נסוגל לעמוד 3 נסוגל לעמוד 3 נסוגל לעמוד 5 נסוגל לשבת 6 נסוגל לעמוד 5 נסוגל לשבת 6 נסוגל לעמוד 6 נסוגל לשבת 6 נסוגל לשבת 6 נסוגל לשבת 6 נסוגל לשבת 6 נסוגל לעמוד 1 דקה בבטיחות 6 נסוגל לעמוד מוסגל לעמוד 6 נסוגל מלמוד 6 נסוגל לעמ | | | | מסוגל לעמוד עצמאית בעזרת ידיים | 3 |
| עמידה ללא תמיכה : עפור במשך 2 דקות ללא תמיכה | | | | מסוגל לעמוד בעזרת ידיים לאחר מספר ניסיונות | 2 |
| עמידה ללא תמיכה: עמוד במשך 2 דקות ללא תמיכה מיסוגל לעמוד בבטיחות 2 דקות | | | | זקוק לעזרה קלה לעמוד או להתייצב | |
| מסוגל לעמוד בבטיחות 2 דקות משרום מסוגל לעמוד בבטיחות 2 דקות בשרוח מסוגל לעמוד 3 שניות ללא תמיכה מסוגל לעמוד 30 שניות ללא תמיכה זקוק למספר ניסיונות לעמוד 30 שניות ללא תמיכה זקוק למספר ניסיונות לעמוד 30 שניות ללא תמיכה זקוק למספר ניסיונות לעמוד 30 שניות ללא עזרה זקוק למספר ניסיונות לעמוד 30 שניות ללא עזרה מסוגל לשבת בכטיחות למשך 2 דקות מסוגל לשבת 30 שניות 5 דקות מסוגל לשבת 30 שניות 5 דקות מסוגל לשבת 30 שניות 5 דקות מסוגל לשבת 30 שניות 5 דקות מסוגל לשבת 40 שניות 5 דקות מסוגל לשבת 50 שניות 5 דקות מסוגל לשבת 40 שניות 5 דקות מסוגל לשבת 50 שניות מסוגל לשבת 50 שניות 5 דקות 6 שניות 5 דקות 6 דקות 6 | | | | זקוק לעזרה בינונית או מרבית לעמוד | |
| מסוגל לעמוד 2 דקות בהשגחה 2 מסוגל לעמוד 3 שניות ללא תמיכה 3 מסוגל לעמוד 30 שניות ללא תמיכה 4 זקוק למספר ניסיונות לעמוד 30 שניות ללא תמיכה 5 מינו מסוגל לעמוד 30 שניות ללא עזרה 6 מינו מסוגל לשבוד 30 שניות ללא עזרה 7 מסוגל לשבת בבטיחות למשך 2 דקות 8 מסוגל לשבת בבטיחות למשך 2 דקות 9 מסוגל לשבת בחשגחה 2 דקות 1 מסוגל לשבת 30 שניות 1 מסוגל לשבת 10 שניות 9 מסוגל לשבת 10 שניות 1 מסוגל לשבת 10 שניות 9 אינו מסוגל לשבת ללא תמיכה 10 שניות 1 מסוגל לשבת ליד מנימלית של ידיים 8 יישב בבטיחות עם עזרה מינימלית של ידיים 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 1 מתיימים לבד אך לא שלט בירידה 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 1 מתיימים לבד אך לא שלט בירידה 9 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 1 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 1 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור בבטיחות עם עזרה מינימלית אל ידיים 1 מסוגל לעבור בבטיחות עם עזרה מינימלית אל ידיים 9 מסוגל לעבור בבטיחות עם עזרה מינימלית אל ידיים 1 מסוגל לעבור שם הוראות מילוליות ו/ או השגחה 9 מסוגל לעבוד 10 שניות בבטיחות 9 מסוגל לעבוד 10 שניות בבטיחות 1 מסוגל לענוד 10 שניות בבטיחות 9 מסוגל לענוד 10 שניות בבטיחות 1 מיני מסוגל לענוד 10 שניות בטיחות 1 מסוגל לעצום ענינים 3 שנות אך עשאר יציב 1 מסוגל למצום עלינים באופן עצמאי ולענוד 1 דקה בהשחה 9 מסוגל לתצמד באולים באופן עצמאי ולענוד 1 דקה בהשמחה 9 מסוגל לתצמד בגלים באופן עצמאי ולענוד 1 דקה בהשחחה 9 מסוגל לתצמד בגלים באופן עצמאי ולענוד 1 דקה במשחות | | | | עמידה ללא תמיכה: עמוד במשך 2 דקות ללא תמיכה | 2 |
| מוסוגל לעמוד 30 שניות ללא תמיכה | | | | מסוגל לעמוד בבטיחות 2 דקות | |
| 1 זקוק לנוסבר ניסיונות לעמוד 30 שניות ללא תמיכה 2 אינו מסוגל לעמוד 30 שניות ללא עזרה 3 ישיבה ללא תמיכה, רגליים על הרצפה: שב בשילוב ידיים למשך 2 דקות 4 מסוגל לשבת במטיחות למשך 2 דקות 5 מוסוגל לשבת במטיחות למשך 2 דקות 6 מוסוגל לשבת 60 שניות 7 מוסוגל לשבת 10 שניות 8 עמידה לשבת 10 שניות 9 אינו מסוגל לשבת ללא תמיכה 10 שניות 9 אינו מסוגל לשבת ללא תמיכה 10 שניות 9 אינו מסוגל לשבת ללא תמיכה 10 שניות 9 אינו מסוגל לשבת ללא תמיכה 10 שניות 9 שולט בישיבה ע"י שימוש בידיים 1 מוחישב לבד אך לא שולט בירידה 9 מוחישב לבד אך לא שולט בירידה 1 מוחישב לבד אך לא שולט בירידה 9 מוחיב לעורה בישיבה 1 מוחיב לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מוחגל לעבור בבטיחות עם עזרה מינימלית של ידיים 1 מוחגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מוחגל לעבור בבטיחות עם עזרה מינימלית של ידיים 1 זקוק לאדם אחד לעזרה 9 מוחגל לעבור בבטיחות עם שורה ממשית של ידיים 1 זקוק לאדם אחד לעזרה 9 מוחגל לעבור בבטיחות עם עזרה מינימלית או או השגחה 1 זקוק לאדם אחד לעזרה 9 עמידה ללא תמיכה עם עינים עצומות: עצום את עיניך ועמוד ישר במשך 10 שניות עם השגחה 1 אינו מוסוגל לעמוד 10 שניות עם השגחה 1 אינו מוסוגל לעמוד 10 שניות כם השגחה 1 אינו מוסוגל לעמוד 10 שניים 3 שניות אך נשאר יציב מוסוגל לתצום עניים 3 שניות אך נשאר יציב מוסוגל לתצומי דר לליים באופן עצמאי ולעמוד 1 דקה במשרחה 7 עמידה ללא תמיכה עם דגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל להצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל להצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל להצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל לתצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל להצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל להצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל לתצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל לתצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסיבה מוסוגל לתצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסוגל לתצמיד הגליים באופן עצמאי ולעמוד 1 דקה במשרחה מוסיבה מוס בת במשרחה מוס במול במשרחה מוסיבה במשרחה מוסיבה במשרחה מוסיבה במשרחה מוסיבה במשרחה מוסיבה במשרחה מוסיבה במשרחה מוסיבה במוד מוסיבה במשרחה מוסיבה במשרחה מוסיבה במוס במוס במידה במוסיבה במוס במוס במוס במוס במ | | | | מסוגל לעמוד 2 דקות בהשגחה | |
| אינו מסוגל לעמוד 30 שניות ללא עזרה | | | | | |
| ישיבה ללא תמיכה, רגליים על הרצפה: שב בשילוב ידיים למשך 2 דקות מסוגל לשבת בבטיחות למשך 2 דקות מסוגל לשבת 6 שניות מסוגל לשבת 6 שניות מסוגל לשבת 10 שניות עמידה לשיבה: שב בבקשה עמידה לשיבה: שב בבקשה עמידה לשיבה: שב בבקשה עמידה לשיבה: שב בבקשה עמידה לשיבה מייי שימוש בידיים מעותה מערים: עבור ברגלים כנגד הכיסא לשליטה בישיבה משעמת) מעברים: עבור בבקשה מהכיסא לשמיטה ובחזרה. (לכיון כיסא עם משעמת, ולכיון כיסא ללא מסוגל לעבור בבטיחות עם עזרה מנינימלית של ידיים מטוגל לעבור בבטיחות עם עזרה מנינימלית של ידיים מטוגל לעבור בבטיחות עם עזרה מנינימלית של ידיים מוסוגל לעבור בבטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בבטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בבטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בבטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בטיחות עם עזרה מנישית של ידיים מוסוגל לעבור בטיחות עם עזרה מנישית של ידיים מוסוגל לעבור מה הראות מילוליות ו/ או השגחה מוסוגל לעמוד 10 שניות בטיחות מוסוגל לעמוד 10 שניות בטיחות מוסוגל לעמוד 10 שניות בטיחות מוסוגל לעמוד 10 שניות בטיחות מוסוגל לעמוד 3 שניות עם השגחה עמידה ללא תמיכה עם רגליים צמודות: הצמד את רגלין ועמוד ללא תמיכה מוסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות עמידה ללא תמיכה עם רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מוסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מוסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מוסוגל להצמיד רגליים באופן עצמאי אן אינו מסוגל לעמוד 2 מוסוגל להצמיד רגליים באופן עצמאי אן אינו מסוגל לעמוד 2 מוסוגל להצמיד רגליים באופן עצמאי אן אינו מסוגל לעמוד 2 מוסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות | | | | | |
| 4 מסוגל לשבת בבטיחות למשך 2 דקות 2 מסוגל לשבת 6 שניות 3 מסוגל לשבת 60 שניות 1 מסוגל לשבת 60 שניות 5 מסוגל לשבת 60 שניות 6 מסוגל לשבת 61 שניות 7 עמידה לשיבה: שב בבקשה 8 יישב בבטיחות עם עזרה מינימלית של ידיים 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 1 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 1 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 6 משנת בל בדא דץ לא שולט בירידה 7 משעות) 5 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 8 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 1 זקוק לאדם אחד לעזרה 9 מסוגל לעבור בטיחות צס עזרה מושית של ידיים 1 זקוק לאדם אחד לעזרה 6 מסוגל לעבור צם הוראות בילוליות ו/ או השגחה 6 עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות בסיחות בסיחות עם יניה שגמה 6 מסוגל לעמוד 10 שניות בבטיחות 7 עמידה ללא תמיכה עם עיניים צמודות:הצמד את רגליך ועמוד ללא תמיכה לוניעת נפילה 9 וקוק לעזרה למניעת נפילה 9 מסוגל לתצום עיניים באופן עצמאי ולעמוד 1 דקה בבטיחות 7 עמידה ללא המיכה עם רגליים באופן עצמאי ולעמוד 1 דקה במטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשרח במשך 60 שניות בליים באופן עצמאי ולעמוד 1 דקה במשחת במשך 20 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשחת במשות במשות במיחות במסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשחת במשך 30 שניות במיחות במסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשחת במשרמת במיד רגליים באופן עצמאי ולעמוד 1 דקה במשחת במשרמת במוגל לתצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשחת במשרת במיחות באומן עצמאי ולעמוד 1 דקה במיחות במיחות במיחות במיחות באומן עצמאי ולעמוד 1 דקה במיחות במיחו | | | | אינו מסוגל לעמוד 30 שניות ללא עזרה | |
| מסוגל לשבת בהשגחה 2 דקות מסוגל לשבת 30 שניות מסוגל לשבת 10 שניות מסוגל לשבת 10 שניות אינו מסוגל לשבת 10 שניות <b>4</b> עמידה לישיבה בבקשה אינו בטיחות עם עזרה מינימלית של ידיים משתמש בגב בהגלים כנגד הכיסא לשליטה בישיבה מערמים בגב הרגלים כנגד הכיסא לשליטה בישיבה מערמים בגב הרגלים כנגד הכיסא לשליטה בישיבה מערמים בישיבה מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בטיחות עם עזרה מימשית של ידיים מסוגל לעבור בטיחות עם עזרה מילוליות ו/ או השגחה מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות עם השגחה מסוגל לעמוד 10 שניות אך נשאר יציב מסוגל לעמוד 10 שניות באום אות אך נשאר יציב מסוגל לעמוד 10 שניות בשיחות מסוגל לעמוד 10 שניות באום אות הצמד את רגלין ועמוד ללא תמיכה עם רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל לתצמיד רגליים באופן עצמאי ולעמוד 1 דקה במטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשרח במשך 30 שניות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשרח במשך 30 שניות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשרח במשך 30 שניות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה במשרח במשך 30 שניות | | | | ישיבה ללא תמיכה, רגליים על הרצפה: שב בשילוב ידיים למשך 2 דקות | |
| 2 מסוגל לשבת 30 שניות 1 מסוגל לשבת 10 שניות 2 אינו מסוגל לשבת 10 שניות 5 אינו מסוגל לשבת 10 שניות 6 אינו מסוגל לשבת 10 שניות 7 עמידה לישיבה: שב בבקשה 8 יושב בבטיחות עם עזרה מינימלית של ידיים 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 1 מתיישב לבד אך לא שולט בירידה 9 זקוק לעזרה בישיבה 5 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 6 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 7 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור בבטיחות עם עזרה מישימת של ידיים 1 זקוק לאדם אחד לעזרה 9 נמסוגל לעבור בטיחות עם עיניים עצומות: עצום את עיניך ועמוד ישר במשך 10שניות בטיחות 9 עמידה לא תמיכה עם עיניים עצומות: עצום את עיניך ועמוד ישר במשך 10שניות שם השגחה 9 מסוגל לעמוד 10 שניות בבטיחות 1 מסוגל לעמוד 10 שניות שם השגחה 1 מסוגל לעמוד 10 שניות שם השגחה 1 אינו מסוגל לעצוד 6 שניות אך נשאר יציב 1 זקוק לעזרה למניית נפילה 1 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 1 זקוק לעזרה למניית נפילה 1 מסוגל לעצום ד 10 שניות בו אובן עצמאי ולעמוד 1 דקה בבטיחות 9 זקוק לעזרה למניית נפילה 1 מסוגל להצמיד רגליים באובן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באובן עצמאי ולעמוד 1 דקה בבטיחות 2 מסוגל להצמיד רגלים באובן עצמאי ולעמוד 1 דקה בבטיחות | | | | מסוגל לשבת בבטיחות למשך 2 דקות | 4 |
| 1 מסוגל לשבת 10 שניות 4 עמידה לשבת ללא תמיכה 10 שניות 5 עמידה לישיבה: שב בבקשה 6 יושב בבטיחות עם עזרה מינימלית של ידיים 7 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 8 שולט בישיבה עייי שימוש בידיים 9 משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה 9 זקן לעזרה בישיבה 1 מתיישב לבד אך לא שולט בירידה 6 משעמת) 5 משעמת) 6 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור בבטיחות עם עזרה מינשית של ידיים 1 זקוק לאדם אחד לעזרה 9 מסוגל לעבור בטיחות עם עזרה מינימלית של ידיים 1 זקוק לאדם אחד לעזרה 6 מסוגל לעבור עם הוראות מילוליות ו/ או השגחה 7 מסוגל לעמוד 10 שניות בבטיחות 8 מסוגל לעמוד 10 שניות שם הוראות בישים עזרח מושות: עצום את עיניך ועמוד ישר במשך 10שניות בטיחות 9 עמידה ללא תמיכה עם עיניים עצומות: עצום את עיניך ועמוד לשר במשך 10שניות עם השגחה 1 מסוגל לעמוד 10 שניות שם השגחה 9 מסוגל לעמוד 10 שניות שם השגחה 1 אינו מסוגל לעמוד 3 שניות ב שניות אך נשאר יציב 9 מסוגל לעמוד 3 שניות 2 שניות אך נשאר יציב 1 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 9 זקוק לעזרה למניעת נפילה 9 עמידה ללא תמיכה עם רגליים צמודות: הצמד את רגליך ועמוד ללא תמיכה עם רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 9 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 10 שניות 2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 10 שניות | | | | מסוגל לשבת בהשגחה 2 דקות | |
| אינו מסוגל לשבת ללא תמיכה 10 שניות | | | | | |
| <ul> <li>י ושב בבטיחות עם עזרה מינינינולית של ידיים</li> <li>שולט בישיבה ע"י שימוש בידיים</li> <li>משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה</li> <li>מתישב לבד אך לא שולט בירידה</li> <li>מקברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא</li> <li>משענות)</li> <li>משענות)</li> <li>מסוגל לעבור בבטיחות עם עזרה מינינולית של ידיים</li> <li>מסוגל לעבור עם הוראות מילוליות ו/ או השגחה</li> <li>זקוק לאדם אחד לעזרה</li> <li>יקוק לאדם אחד לעזרה</li> <li>עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות</li> <li>מסוגל לעמוד 10 שניות עם השגחה</li> <li>מסוגל לעמוד 10 שניות עם השגחה</li> <li>מסוגל לעמוד 3 שניות עם השגחה</li> <li>מסוגל לעמוד 5 שניות</li> <li>מסוגל לעמוד 5 שניות אך נשאר יציב</li> <li>עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה</li> <li>אינו מסוגל לעצום עיניים 3 שנות אך נשאר יציב</li> <li>עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה</li> <li>עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה</li> <li>מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות</li> <li>מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה</li> <li>מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות</li> <li>מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות</li> </ul> | | | | אינו מסוגל לשבת ללא תמיכה 10 שניות | 0 |
| משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה מייי שימוש בידיים משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה מתיישב לבד אך לא שולט בירידה מקיק לעזרה בישיבה מקברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא משענות) מענות) מענות לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מישית של ידיים מסוגל לעבור עם הוראות מילוליות ו/ או השגחה מסוגל לעבור עם הוראות מילוליות ו/ או השגחה מסוגל לעבור או השגחת 2 אנשים עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות עם השגחה מסוגל לעמוד 3 שניות אך נשאר יציב עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה עם רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות עמידה ללא תמיכה עם רגליים באופן עצמאי ולעמוד 1 דקה בהשחחה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשחחה | | | | <b>עמידה לישיבה:</b> שב בבקשה | 4 |
| משתמש בגב הרגלים כנגד הכיסא לשליטה בישיבה מתיישב לבד אך לא שולט בירידה מעברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא משענות) מטוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מומשית של ידיים מסוגל לעבור עם הוראות מילוליות ו/ או השגחה מיקוק לאדם אחד לעזרה עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות מסוגל לעמוד 10 שניות בבטיחות מוסוגל לעמוד 10 שניות בבטיחות מוסוגל לעמוד 10 שניות אך נשאר יציב מוסוגל לעמוד 10 שניות אך נשאר יציב עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | יושב בבטיחות עם עזרה מינימלית של ידיים | |
| 1 מתיישב לבד אך לא שולט בירידה 5 מעברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא 6 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 7 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 8 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 9 מסוגל לעבור עם הוראות מילוליות ו/ או השגחה 1 זקוק לאדם אחד לעזרה 1 זקוק לאדם אחד לעזרה 6 עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות 5 מסוגל לעמוד 10 שניות בבטיחות 7 מסוגל לעמוד 10 שניות אך נשאר יציב 9 מסוגל לעמוד עם השגחה 1 אינו מסוגל לעמוד משניים 3 שניות אך נשאר יציב 1 מסוגל לעצום עיניים 3 שניות אך נשאר יציב 9 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 9 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | | |
| 1 אקוק לעזרה בישיבה 2 מעברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא משענות) 2 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 3 מסוגל לעבור בבטיחות עם עזרה מימשית של ידיים 2 מסוגל לעבור בבטיחות עם עזרה מימשית של ידיים 3 מסוגל לעבור עם הוראות מילוליות ו/ או השגחה 3 וקוק לאדם אחד לעזרה 3 וקוק לאדם אחד לעזרה 4 מסוגל לעמוד מו שניים אנשים 4 מסוגל לעמוד 10 שניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות 4 מסוגל לעמוד 10 שניות בבטיחות 5 מסוגל לעמוד 10 שניות עם השגחה 5 מסוגל לעמוד 10 שניות עם השגחה 5 מסוגל לעמוד 3 שניים 3 שניים 5 שניות אך נשאר יציב 5 מסוגל להצמיד הלא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשתחה 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשתחה 5 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לממוד במשך 30 שניות 5 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות 5 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות 5 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות 5 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| מעברים: עבור בבקשה מהכיסא למיטה ובחזרה. (לכיוון כיסא עם משענות, ולכיוון כיסא ללא משענות) מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים מסוגל לעבור בבטיחות עם עזרה מומשית של ידיים מסוגל לעבור עם הוראות מילוליות ו/ או השגחה זקוק לאדם אחד לעזרה זקוק לאדם אחד לעזרה מסוגל לעמוד מו שניניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות עם השגחה מסוגל לעמוד 3 שניים 3 שניות אך נשאך יציב מסוגל לעמוד 3 שניים 3 שניות אך נשאך יציב מסוגל להצמיד הלא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | · | |
| משעות) 4 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 5 מסוגל לעבור בבטיחות עם עזרה מינימלית של ידיים 6 מסוגל לעבור עם הוראות מילוליות ו/ או השגחה 7 זקוק לאדם אחד לעזרה 6 מסוגל לעמוד 10 שניים עצומות: עצום את עיניך ועמוד ישר במשך 10שניות 8 מסוגל לעמוד 10 שניים עצומות: עצום את עיניך ועמוד ישר במשך 10שניות 9 מסוגל לעמוד 10 שניות בבטיחות 1 מסוגל לעמוד 10 שניות עם השגחה 2 מסוגל לעמוד 10 שניות אך נשאר יציב 1 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 9 זקוק לעזרה למניעת נפילה 9 עמידה ללא תמיכה עם רגליים צמודות: הצמד את רגליך ועמוד ללא תמיכה 9 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 1 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | | 0 |
| מסוגל לעבור בבטיחות עם עזרה ממשית של ידיים מסוגל לעבור עם הוראות מילוליות ו/ או השגחה זקוק לאדם אחד לעזרה מסוגל לעבור או השגחת 2 אנשים מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות בבטיחות מסוגל לעמוד 10 שניות עם השגחה מסוגל לעמוד 10 שניות עם השגחה מסוגל לעמוד 3 שניים זשניות עם השגחה מסוגל לעמוד 3 שניים 3 שניות אך נשאר יציב מסוגל לעצום עיניים 3 שניות אך נשאר יציב מסוגל לעזרה למניעת נפילה עמידה ללא תמיכה עם רגליים צמודות: הצמד את רגליך ועמוד ללא תמיכה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | משענות) | |
| 2 מסוגל לעבור עם הוראות מילוליות ו/ או השגחה 1 זקוק לאדם אחד לעזרה 0 זקוק לעזרת או השגחת 2 אנשים 6 עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות 4 מסוגל לעמוד 10 שניות בבטיחות 5 מסוגל לעמוד 10 שניות עם השגחה 6 מסוגל לעמוד 1 שניות עם השגחה 7 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 0 זקוק לעזרה למניעת נפילה 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 6 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| 1 זקוק לאדם אחד לעזרה 0 זקוק לעזרת או השגחת 2 אנשים 6 עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות 4 מסוגל לעמוד 10 שניות בבטיחות 5 מסוגל לעמוד 10 שניות עם השגחה 6 מסוגל לעמוד 10 שניות עם השגחה 7 אינו מסוגל לעמוד 3 שניית 5 שניות אך נשאר יציב 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 7 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | | |
| 0 זקוק לעזרת או השגחת 2 אנשים 2 עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות 4 מסוגל לעמוד 10 שניות בבטיחות 5 מסוגל לעמוד 10 שניות עם השגחה 6 מסוגל לעמוד 10 שניות עם השגחה 7 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 9 זקוק לעזרה למניעת נפילה 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 7 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה | | | | | |
| <ul> <li>עמידה ללא תמיכה עם עיניים עצומות:עצום את עיניך ועמוד ישר במשך 10שניות</li> <li>מסוגל לעמוד 10 שניות בבטיחות</li> <li>מסוגל לעמוד 10 שניות עם השגחה</li> <li>מסוגל לעמוד 3 שניות עם השגחה</li> <li>אינו מסוגל לעמוד 3 שניות אך נשאר יציב</li> <li>זקוק לעזרה למניעת נפילה</li> <li>עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה</li> <li>מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות</li> <li>מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה</li> <li>מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות</li> <li>מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות</li> </ul> | | | | | |
| 4 מסוגל לעמוד 10 שניות בבטיחות 3 מסוגל לעמוד 10 שניות עם השגחה 4 מסוגל לעמוד 10 שניות עם השגחה 5 מסוגל לעמוד 3 שניות 6 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב 6 זקוק לעזרה למניעת נפילה 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד 2 שניות | | | | | |
| 3 מסוגל לעמוד 10 שניות עם השגחה<br>2 מסוגל לעמוד 3 שניות<br>1 אינו מסוגל לעצום עיניים 3 שניות אך נשאך יציב<br>5 זקוק לעזרה למניעת נפילה<br>7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה<br>4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות<br>5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה<br>6 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד 2 שניות | | | | | |
| 2 מסוגל לעמוד 3 שניות 1 אינו מסוגל לעמוד 5 שניות 8 שניות 1 שניות 7 מסוגל לעצום עיניים 3 שניות אך נשאר יציב 0 זקוק לעזרה למניעת נפילה 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| 1 אינו מסוגל לעצום עיניים 3 שניות אך נשאר יציב<br>0 זקוק לעזרה למניעת נפילה<br>7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה<br>4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות<br>5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה<br>2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| 0 זקוק לעזרה למניעת נפילה 7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות 5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 6 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה 7 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| <ul> <li>7 עמידה ללא תמיכה עם רגליים צמודות:הצמד את רגליך ועמוד ללא תמיכה</li> <li>4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות</li> <li>5 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה</li> <li>2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות</li> </ul> | | | | • | |
| 4 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בבטיחות<br>3 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה<br>2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| 3 מסוגל להצמיד רגליים באופן עצמאי ולעמוד 1 דקה בהשגחה<br>2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | · | - |
| 2 מסוגל להצמיד רגליים באופן עצמאי אך אינו מסוגל לעמוד במשך 30 שניות | | | | | |
| | | | | · | |
| ו אוין לעוון בעבויון בובא אן בוסוגל לעבור כב סביונ עם ואיים בפורו ו | | | | | |
| 0 זקוק לזרה בעמידת מוצא ואינו מסוגל לעמוד 15 שניות | | | | · | |





# המשך -Berg Balance Scale

| 8 | שליחת יד לפנים <b>functional reach:</b> הרם יד ל – 90 מעלות מתח את האצבעות ונסה<br>להגיע לפנים כמה שיותר.(מודדים את ההפרש בין נקודת ההתחלה לסיום).אין לגעת בקיר | תאריך<br>(1) | תאריך<br>(2) | תאריך<br>(3) |
|---|---|---|---|---|
| 4 | יכול להגיע קדימה בבטיחות 25 ס"מ ויותר | | | |
| 3 | יכול להגיע קדימה 12.5 ס"מ בבטיחות | | | |
| 2 | יכול להגיע קדימה 5 ס"מ בבטיחות | | | |
| 1 | מתכופף קדימה אך זקוק להשגחה | | | |
| 0 | זקוק לעזרה למניעת נפילה | | | |
| 9 | הרמת חפץ מהרצפה: עמוד והרם את המעל הנמצאת לפניך | | | |
| 4 | יכול להרים בבטיחות ובקלות | | | |
| 3 | יכול להרים אך זקוק להשגחה | | | |
| 2 | אינו מסוגל להרים אך מגיע למרחק של 2-5 סיימ ושומר על שיימ באופן עצמאי | | | |
| 1 | אינו מסוגל להרים וזקוק להשגחה בזמן הניסיון. | | | |
| 0 | אינו מסוגל לנסות, דורש עזרה למניעת נפילה | | | |
| 10 | הסתובב להסתכל מאחוריך, מעבר לכתף ימין, ושמאל | | | |
| | הסתובב להביט לאחור מעבר לכתף שמאל. חזור שנית מעבר לכתף ימין | | | |
| 4 | מביט לאחור דרך 2 הצדדים ומעביר משקל טוב | | | |
| 3 | מסתובב לאחור לצד אחד טוב. צד שני אינו מעביר משקל היטב | | | |
| 2 | מסתובב לצדדים בלבד אך שומר על יציבות | | | |
| 1 | זקוק להשגחה בזמן סיבוב לאחור | | | |
| 0 | זקוק לעזרה למניעת איבוד שיווי משקל ונפילה | | | |
| 11 | הסתובב 360° מעלות: בצע סיבוב שלם במקום ועצור. בצע סיבוב לצד השני | | | |
| 4 | מסוגל להסתובב 360° בבטיחות ב-4 שניות ופחות לכל כיוון | | | |
| 3 | מסוגל להסתובב 360° בבטיחות לכיוון אחד בלבד ב-4 שניות ופחות | | | |
| 2 | מסוגל להסתובב 360° בבטיחות אך באיטיות | | | |
| 1 | זקוק להשגחה צמודה או הוראות מילוליות | | | |
| 0 | זקוק לעזרה בזמן הסיבוב | | | |
| 12 | החלפת רגליים על שרפרף: הנח לסירוגין רגלים על שרפרף. המשך עד שכל רגל נגעה<br>בשרפרף 4 פעמים | | | |
| 4 | מסוגל לעמוד באופן עצמאי ולסיים 8 צעדים ב-20 שניות | | | |
| 3 | מסוגל לעמוד באופן עצמאי ולסיים 8 צעדים ב-20 שניות ויותר | | | |
| 2 | מסוגל לסיים 4 צעדים ללא עזרה אך עם השגחה. | | | |
| 1 | מסוגל לסיים 2 צעדים או פחות אך דורש עזרה מינימלית | | | |
| 0 | זקוק לעזרה למניעת נפילה / לא מסוגל לנסות | | | |
| 13 | עמידה ללא תמיכה, רגל אחת לפני השניה Tandem :הנח רגל אחת לפני השנייה.<br>אם אינך יכול, נסה להניח עקב של הרגל הקדמית לפני האצבעות של הרגל האחורית | | | |
| 4 | מסוגל לעמוד עמידת TANDEM באופן עצמאי למשך 30 שניות | | | |
| 3 | מסוגל להניח רגל אחת לפני השניה באופן עצמאי ולעמוד במשך 30 שניות | | | |
| 2 | מסוגל לבצע צעד קטן באופן עצמאי ולעמוד 30 שניות | | | |
| 1 | זקוק לעזרה לביצוע צעד, יכול להחזיק 15 שניות | | | |
| 0 | מאבד שיווי משקל בזמן ביצוע צעד או עמידה | | | |
| 14 | עמידה על רגל אחת עמוד על רגל אחת זמן רב ככל שאתה יכול ללא תמיכה | | | |
| 4 | מסוגל להרים רגל באופן עצמאי ולהחזיק 10 שניות ומעלה | | | |
| 3 | מסוגל להרים רגל באופן עצמאי ולהחזיק 5-10 שניות | | | |
| 2 | מסוגל להרים רגל באופן עצמאי ולהחזיק 3-5 שניות | | | |
| 1 | מנסה להרים רגל. אינו מסוגל להחזיק 3 שניות אך נשאר עומד באופן עצמאי | | | |
| 0 | אינו מסוגל לנסות או זקוק לתמיכה למניעת נפילה | | | |
| | ציון סופי: | 1 | | |







### :ארגון הסביבה

מסלול של 10 מטרים מסומן ע"י שני קוים. כסא מונח שני מטרים אחרי קו סוף המסלול.

#### <u>עמדת מוצא</u>:

נבדק עומד שני מטרים לפני תחילת המסלול.

### ההוראה שיש לתת לנבדק:

לך ישר קדימה במהירות הנוחה לך, בלי להאט או לעצור, עד לכסא שבקצה המסלול.

#### אופן ביצוע המדידה:

התחל את המדידה עם סטופר כשהנבדק חוצה את קו תחילת המסלול. עצור את המדידה כשהנבדק חוצה את קו סוף המסלול.

בנוסף למדידת המהירות ספור את מספר הצעדים שמבצע הנבדק מרגע הפעלת הסטופר עד עצירתו.

### משתנים נורמליים של הליכה

מהירות הליכה למרחקים קצרים:

| 70 | 60 | 50 | 40 | 30 | עשור |
|---|---|---|---|---|---|
| הליכה במהירות הנוחה (מטר/שניה) | | | | | |
| 1.33 | 1.37 | 1.47 | 1.47 | גברים | |
| 1.26 | 1.3 | 1.4 | 1.4 | 1.42 | נשים |
| הליכה במהירות המקסימלית (מטר/שניה) | | | | | |
| 2.08 | 1.93 | 2.1 | 2.47 | 2.45 | גברים |
| 1.75 | 1.76 | 2 | 2.12 | 2.5 | נשים |

:מתוך

Bohannon RW. Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants. Age and Ageing 1997; 26: 15-19

1.87 : Cadence צעדים בדקה 112 צעדים בדקה אורך צעד: 0.72 מטר

### סיווג הליכה לפי מהירות ההליכה

0.16-0.25 m/sec הבית: מחגבלת במסגרת הבית: 0.26-0.42 m/sec הליכה ללא הגבלה בבית: 0.43-0.79 m/sec הליכה מוגבלת בקהילה: מיטית: 0.8-1.2 m/sec הליכה לא מוגבלת בקהילה, איטית: 0.8-1.2 m/sec

מבוסס על: Peny J





# Six minute walk

המבתן מיועד לבדיקת סיבולת הליכה.

הציוד הנדרש הינו שעון עצר ומרחק הליכה מדוד.

### הנחיות לנבדק:

הנבדק עומד בתחילת המסלול. ההנחיה הניתנת "לך כמה שיותר מהר למשך 6 דקות על מנת לעבור את המרחק הגדול ביותר. אתה יכול לעצור במידה ואתה זקוק אך נסה להמשיך ברגע שאתה מסוגל."

#### הנחיות לבודק:

עם תחילת ההליכה מופעל שעון העצר ובתום 6 דקות הנבדק מתבקש לעצור. הבודק מחשב את מרחק ההליכה שהושג. על הבודק להמנע מעידוד הנבדק במהלך המבחן. ניתן לידע על הזמן שנישאר לאחר 2 ו4 דקות.

יש לאפשר לנבדק לעצור ולעמוד או לשבת במידה והוא זקוק לכך. זמן המנוחה כלול בזמן המבחן.

(Butland et al, 1982; Guyatt et al, 1985)

### משתנים נורמלים עבור נבדקים בריאים:

| גברים מרחק ממוצע | נשים מרחק ממוצע | גיל |
|----------------------|----------------------|-------|
| 800 <u>+</u> 83 מטר | 37 <u>+</u> 699 מטר | 20-40 |
| מטר 56 <u>+</u> 671 | 85 <u>+</u> 670 מטר | 41-60 |
| 89 <u>+</u> 687 פמטר | 583 <u>+</u> 583 מטר | 61-80 |

(Gibbons et al, 2001)

### משתנים נורמלים עבור קשישים בקהילה:

| גברים מרחק ממוצע | נשים מרחק ממוצע | גיל |
|---------------------|---------------------|-------|
| 92 <u>+</u> 572 מטר | 92 <u>+</u> 538 מטר | 60-69 |
| 85 <u>+</u> 527 מטר | מטר 75 <u>+</u> 471 | 70-79 |
| 73 <u>+</u> 417 מטר | 85 <u>+</u> 392 מטר | 80-89 |

(Steffen et al, 2002)

# **ACTIVITIES-SPECIFIC BALANCE CONFIDENCE (ABC) SCALE**

אנא ציין את מידת הביטחון שלך לבצע את הפעולות הבאות מבלי לאבד שיווי משקל על ידי ציון האחוז בסקאלה מ 0% עד 100%.

אם אינך מבצע כיום את הפעילות שבשאלה, נסה לדמיין עד כמה בטוח היית אילו היית מבצע אותן.

אם הנך נעזר באביזר עזר להליכה אנא דרג את רמת הביטחון שלך כשאתה משתמש באביזר זה.

| 0% | 10 | 20 | 30 | 40 | 50 | 60 | 70 | 80 | 90 | 100% | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| לא<br>בטוח | | | | | | | | | | בטוח<br>לחלוטין | |
| | | נה | אשר אר: | א יציב כ | תהיה ל | ושקל או | שיווי מ | א תאבד | טוח של: | מה הנך ב: | עד כ |
| | | | | | | | _ % | ך הבית | זלך בתו | 1מתו | |
| | | | | | | | _ % | מדרגות: | ז ויורד ב | 2עולו | <u> </u> |
| | | | | | % | רצפה | בית מר | רים נעל | ופף להו: | 3מתכ | } |
| | | _ | | % | עיניים | כגובה הי | למדף ב | י להגיע | יט יד כד | 4מוש | ļ |
| | | ַנות % | נ האצבע | על קצור | ך עומד: | אשר הנ: | למדף כ | י להגיע | יט יד כד | 5מוש | ; |
| | | | _ % ? | על כיסא | ך עומד: | אשר הנ: | למדף כ | י להגיע | יט יד כד | 6מוש | ; |
| | | | | | | | _ % | הרצפה | וטא את | 7מטא | , |
| | | | | _ % i | ה בחניה | ית החונ | אל מכונ | ץ לבית א | זלך מחו | 8מתו | } |
| | | | | | | | % | מכונית | יוצא מו/י | 9נכנכ | ) |
| | | | | | _ | | % | חניה | ה מגרש | 10חוצו | ) |
| | | | | % (ה | פע (רמפ | טח משונ | רד משנ | ז או במו | במעלו ב | 11הולן | |
| | | % : | במהירות | ל פניך נ | וולפים ע | אנשים ר | רם, כשי | הומה אז | בקניון | 12הולן | <u> </u> |
| | | | | | 9 | אבך %' | ם נתקל | קניון ואד | בתוך ז | 13הולן | } |
| | | | % | עקה מׁ | ויזה במי | תוך אר: | ות נעות | במדרג - | ז או יורז | 14עולו | 1 |
| | | | % | עקה מ | ויזה במי | ללא אר: | ות נעות | במדרג ٔ | ז או יורז | 15עולו | ; |
| | | | | _ | | % | קרח | רכה עם | על מד | 16הולן | ) |

Powell LE & Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol Med Sci 1995; 50 (1):M28-34